CLINICAL TRIAL: NCT06698562
Title: Effect of Virtual Reality and Laser Biostimulation on Pain Perception and Dental Anxiety in Children
Brief Title: Virtual Reality and Laser Biostimulation on Pain Perception and Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SIRIN GUNER ONUR (Other)
Responsible Party: Sponsor-Investigator, SIRIN GUNER ONUR, Associate Professor, Altinbas University
Organization: Altinbas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/143
Record Dates: First submitted 2024-11-15; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Dental Anxiety; Pain Intensity Assessment
Keywords: pain perception; dental anxiety; children; virtual reality; dental laser
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: The study included 40 Frankl "positive" and "definitely positive" pediatric patients between the ages of 6 and 10, applied to Altinbaş University Faculty of Dentistry Pediatric Dentistry Clinic for routine dental treatments between January 2023 and April 2023, and had no previous local anesthesia experience.
  This study designed as a randomized, single-center, split-mouth, double blind clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group IIa Tell- Show-Do (Active Comparator): Placebo topical anesthesia + LLLT + Local anesthesia
  Interventions: Other: Tell Show Do Group + LLLT; Other: Tell Show Do Group
- Group IIb Tell- Show-Do (Placebo Comparator): Topical anesthesia + placebo LLLT + Local anesthesia
  Interventions: Other: Tell Show Do Group
- Group Ia Distraction (VR) (Active Comparator): Placebo topical anesthesia + LLLT + Local anesthesia
  Interventions: Other: Distraction with Virtual reality glassess + LLLT
- Grup Ib Distraction (VR) (Placebo Comparator): Topical anesthesia + placebo LLLT + Local anesthesia
  Interventions: Other: Distraction with Virtual reality glassess

INTERVENTIONS:
Other: Distraction with Virtual reality glassess — the injection site was dried with a cotton pellet and placebo topical anaesthesia was applied with a pre-sterilised wooden ear stick in a circular motion followed by laser biostimulation. The Wiser diode laser (Doctor Smile, Vicenza, Italy), a diode laser device with a wavelength of 980 nm and equipped with a 600 μm diameter fibre, was used to deliver low-level laser therapy to the area of interest. The tip of the laser carrier system was placed at a distance of 1 cm from the target tissue without contact and applied with continuous circular movements as recommended by the manufacturer. A silicone piece was placed on the end of the carrier system to ensure that the distance to the tissue remained constant in each application. The focal spot area was determined as 0.087 cm2. The power of the laser used in our study was determined as 0.3 W and the application time was selected as 60 seconds. The patient and the physician wore protective goggles during the whole procedure to prevent possi
  Arms: Grup Ib Distraction (VR)
Other: Distraction with Virtual reality glassess + LLLT — The injection area was dried with a cotton pellet before injection. A topical anaesthetic gel containing 20% benzocaine (Vision pat gel) was applied to the mucosal tissues to be injected using a pre-sterilised ear stick. After the application of the topical anaesthetic agent, the laser device was positioned in the same way, but without applying energy, and the sound of the laser device was pre-recorded and the study was blinded. In this way, a placebo effect was created and the patient was prevented from distinguishing between the laser and non-laser session. After this procedure, local anaesthesia was applied.
  Arms: Group Ia Distraction (VR)
Other: Tell Show Do Group + LLLT — The injection site was dried with a cotton pellet and placebo topical anaesthesia was applied with a pre-sterilised wooden ear stick in a circular motion followed by laser biostimulation. The Wiser diode laser (Doctor Smile, Vicenza, Italy), a diode laser device with a wavelength of 980 nm and equipped with a 600 μm diameter fibre, was used to deliver low-level laser therapy to the area of interest. The tip of the laser carrier system was placed at a distance of 1 cm from the target tissue without contact and applied with continuous circular movements as recommended by the manufacturer. A silicone piece was placed on the end of the carrier system to ensure that the distance to the tissue remained constant in each application. The focal spot area was determined as 0.087 cm2. The power of the laser used in our study was determined as 0.3 W and the application time was selected as 60 seconds. During the whole procedure, the patient wore virtual glasses and the physician wore protective go
  Arms: Group IIa Tell- Show-Do
Other: Tell Show Do Group — In this session, the injection area was dried with a cotton pellet before injection. A topical anaesthetic gel containing 20% benzocaine (Vision pat gel) was applied to the mucosal tissues to be injected using a pre-sterilised ear stick. After the application of the topical anaesthetic agent, the laser device was positioned in the same way, but without applying energy, and the sound of the laser device was pre-recorded and the study was blinded. In this way, a placebo effect was created and the patient was prevented from distinguishing between the laser and non-laser session. After this procedure, local anaesthesia was applied.
  Other Names: Group IIb
  Arms: Group IIa Tell- Show-Do; Group IIb Tell- Show-Do

SUMMARY:
Dental anxiety in children can prevent planned treatment from being carried out, negatively affect the child's relationship with the dentist and make the treatment process difficult. The most common sources of directly anticipated anxiety are known to be associated with pain. Painful experiences are anxiety-provoking for people of all ages, especially children.This study aims to evaluate the effect of virtual reality glassess (VR) and low-level laser therapy (LLLT) on dental anxiety and pain perception during local anaesthesia administration in paediatric patients.

DETAILED DESCRIPTION:
This study aims to investigate the combined effects of virtual reality glassess (VR) and low-level laser therapy (LLLT) on dental anxiety and pain perception in paediatric patients undergoing local anaesthesia for dental procedures. Dental anxiety is a common issue in children, often leading to increased pain perception and poor cooperation during treatment. Virtual reality has been proposed as a distraction technique, while LLLT is believed to reduce pain and inflammation. By exploring the effectiveness of these two interventions, the study seeks to determine whether VR and LLLT can serve as effective adjuncts to improve patient comfort, reduce anxiety, and enhance overall treatment experience during the administration of local anaesthesia

ELIGIBILITY:
Inclusion Criteria:

* No history of systemic disease or infectious disease
* Compliant with the dental treatments to be performed in the Children's Dental Hospital and able to answer the questions asked
* Exhibiting 'positive' and 'absolutely positive' behaviours during the examination, compliant according to the Frankl scale,
* Children with no previous experience of dental treatment with local anaesthesia

Exclusion Criteria:

* Children with any systemic condition
* Mentally and physically disabled, unable to co-operate,
* Children allergic to local anaesthesia,
* Previous dental treatment experience with local anaesthesia
* Exhibiting "negative" and "strongly negative" behaviour according to the Frankl scale
* Children with eye diseases such as myopia and astigmatism

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Pain perception | Right before and immediately after treatment
  In this study, each patient received both topical anaesthesia and DSLT treatment using a split-mouth design.Pain perception was measured by Wong and Baker scale. In this scale there are 6 different facial expressions ranging from very happy to very unhappy to express the level of pain.The scale includes six faces, each illustrating a different level of pain intensity:
  0 (No Pain), 1 (Very Mild Pain), 2 (Mild Pain), 3 (Moderate Pain), 4 (Severe Pain) 5 (Very Very Severe Pain). The Wong Baker facial expression pain scale was evaluated right before and immediately after the application of local anesthesia by an observer physician other than the physician administering local anesthesia. The pictures on this scale were introduced to the patient in an appropriate language. Right before and immediately after local anesthetic injection, the picture chosen by the patient was recorded on the scale.
Dental Anxiety | Right before and immediately after treatment
  Dental anxiety levels of the children were physiologically evaluated using the 'Venham Picture Test'. The picture chosen by the patient was recorded on the scale. The Venham Picture Test was assessed right before and immediately after local anaesthetic injection by an observer clinician other than the clinician administering the local anesthesia. The children were shown 8 pairs of pictures of boys (one "anxious" picture and one "non-anxious" picture), each drawn in a contrasting mood, and were asked to choose the picture on each card that corresponded to their feelings. A score of 1 was given if the child chose the "anxious" picture and 0 if the child chose the "non-anxious" picture. To determine the total score, the number of "anxious" pictures was summed (lowest score 0, highest score 8).
Pain perception | During local anesthesia application
  The "Face, Legs, Activity, Cry, Consolability (FLACC)" pain assessment scale was also evaluated during local anesthesia application by an observer clinician other than the clinician to whom local anesthesia would be applied. The patient's reactions were evaluated by observation by the researcher. Pain values were determined between 0-2 for each parameter and 0-10 for the total scale score. According to the scale, the total score was evaluated as follows: 0: No pain, 1-3: Mild pain, 4-6: Moderate pain and discomfort, 7-10: Severe pain and discomfort.

SECONDARY OUTCOMES:
Dental Anxiety | Right before, during and immediately after the application of local anesthesia
  Pulse rate and oxygen saturation values were measured with a pulse oximetry device. The measurement was started by attaching the finger apparatus of the device to the index finger of the left hand of the patients. Then, the pulse and SpO2 values right before, during and immediately after the application of local anesthesia were recorded. At the end of the session, these values were averaged and recorded in the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: SIRIN GUNER ONUR, PhD, Study Director
Locations (1):
- Altinbas University Faculty of Dentistry, Istanbul, Marmara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No